CLINICAL TRIAL: NCT01735097
Title: A Double-blind, Randomized, Placebo-controlled Trial of Nigella Sativa in the Treatment of Palmer Arsenical Keratosis
Brief Title: Effect of Nigella Sativa in the Treatment of Palmer Arsenical Keratosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU-002-CT
Record Dates: First submitted 2012-11-15; First posted 2012-11-28 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Arsenical Keratosis
Keywords: Arsenic; Keratosis; Nigella sativa; Palm; Vitamin E
MeSH Terms: conditions — Keratosis | interventions — Vitamin E; Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arsenical keratosis (Study) (Experimental): Vitamin E (200 mg, soft capsule) plus Nigella sativa (500 mg, soft capsule) twice daily, orally for 12 weeks
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Nigella sativa
- Arsenical keratosis (Control) (Active Comparator): Vitamin E (200 mg, soft capsule) plus Placebo (refined oil in soft capsule with same size and color as that contains N sativa) twice daily, orally for 12 weeks
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin E — Vitamin E (200 mg, soft capsule)
Dietary Supplement: Nigella sativa — Nigella sativa (200 mg, soft capsule)
  Arms: Arsenical keratosis (Study)
Dietary Supplement: Placebo — Placebo (refined oil in soft capsule with same color and size like that contains N. sativa)
  Arms: Arsenical keratosis (Control)

SUMMARY:
Daily intake of Nigella sativa for 12 weeks is effective in the treatment of palmer arsenical keratosis

DETAILED DESCRIPTION:
Depending on inclusion and exclusion criteria total 40 patients of palmer arsenical keratosis patients (both male and female; age range 18- 60 years) will be recruited from an arsenic affected area. Study population will be divided randomly into two equal groups: one group will receive vitamin E capsules (200 mg) plus placebo and another group will receive vitamin E capsule plus N. sativa capsules (500 mg) twice daily for 12 weeks. Drinking water (50 mL) and urine (50 mL) samples will be collected before starting the study and estimate the amount of total arsenic in order to confirm the diagnosis. Nail (approx. 1 g) and blood (5 mL) samples will be collected both before and completion of the study to see the efficacy and safety of the drug. Clinical examinations will be done at regular interval (two weeks). Clinical features and adverse effects will be recorded using a structured data collection sheet. Plasma cholesterol, vitamin E, and total antioxidant, serum transaminase, billirubin, creatinine levels and arsenic level in nail will be measured to evaluate the effectiveness of N. sativa on palmer arsenical keratosis patients

ELIGIBILITY:
Inclusion Criteria:

* Moderate palmer arsenical keratosis
* Patient drinking arsenic contaminated water (more than 0.05 mg/L) for more than six months
* Subjects those voluntarily agree to participate

Exclusion Criteria:

* Patient received treatment of arsenicosis for the last three months
* Pregnancy
* Lactating mother
* Eczema
* Psoriasis
* Contact dermatitis
* Tuberculosis
* Diabetes mellitus
* Patients with hepatic and renal impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of signs and symptoms of palmer arsenical keratosis | up to 12 weeks
  Signs and symptoms of palmer arsenical keratosis will be examined by one trained doctor at the temporary arsenic camp at regular interval (2 weeks). Another doctor will note the findings of the patient in the data collection sheet without informing the previous data to the former doctor.
  Signs and symptoms of moderate arsenical keratosis will be assessed by estimating the number and size of keratotic lesions and expressed into scoring.

SECONDARY OUTCOMES:
Arsenic level in nails | 0 week (baseline), 12 weeks (end)
  Amount of arsenic in nails will be estimated by Atomic Fluorescence spectrometry (AFS) both before and after completion of treatment.
Estimation of serum vitamin E levels | 0 week (baseline), 12 weeks (end)
  To see any change in the concentration of plasma vitamin E levels after use of N.sativa capsules. This parameter will be estimated by spectrophotometric method.
Estimation of serum total cholesterol levels | 0 week (baseline), 12 weeks (end)
  To see any change in the concentration of serum cholesterol levels after use of N. sativa. This parameter will be estimated by spectrophotometric method.
Liver function | 0 week (baseline), 12 weeks (end)
  To see any change in the concentration of serum bilirubin, transaminase levels after use of N. sativa. These parameters will be estimated by spectrophotometric method.
Renal function | 0 week (baseline), 12 weeks (end)
  To see any change in the concentration of blood urea and serum creatinine levels after use of N. sativa. These parameters will be estimated by spectrophotometric method.

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, MBBS, PhD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh